CLINICAL TRIAL: NCT01929824
Title: A Pilot Study: Nasal Nitric Oxide Levels in Eosinophilic Esophagitis.
Brief Title: Nasal Nitric Oxide Levels in Eosinophilic Esophagitis (EoE)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vivek N Iyer, Principal Investigator, Mayo Clinic
Other Study IDs: 13-001194
Record Dates: First submitted 2013-08-14; First posted 2013-08-28 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: dysphagia, trouble swallowing, chest pain
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Oral Nitric Oxide testing — o Oral nitric oxide is measured by a breathing test where the participant will be seated in a chair and asked to breathe out into a small hand-held instrument for about 6 seconds.

SUMMARY:
This study is aimed at understanding whether oral nitric oxide levels can be used as a non-invasive marker for the diagnosis and management of patient with eosinophilic esophagitis (EoE).

DETAILED DESCRIPTION:
Nitric oxide (NO) is produced by activated eosinophils and oral NO levels are known to be elevated in asthma and eosinophilic bronchitis. The measurement of oral NO is a non-invasive,easy to perform low cost procedure that is used frequently in the diagnosis and management of asthma. The diagnosis of eosinophilic esophagitis (EoE) requires conscious sedation, an upper endoscopy with biopsy, and histologic evaluation of the biopsy specimen. This is a costly and somewhat invasive procedure. If oral NO was elevated as a result of activity of esophageal eosinophils in EoE, the measurement of oral NO may potentially be a very convenient and useful test in the evaluation and treatment of EoE. We propose a pilot study to determine if oral NO levels are elevated in patients with eosinophilic esophagitis.

ELIGIBILITY:
Inclusion criteria:

* Subjects with dysphagia and active esophageal infiltration (esophageal eosinophilic count of >/= 15 eos/hpf)
* Subjects with or without a clinical diagnosis of asthma

Exclusion criteria:

* Subjects with chronic cough
* Severe CAD
* MI within the last 3 months
* Cystic fibrosis
* Tuberculosis
* Chronic obstructive pulmonary disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eosinophilic esophagitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Number of patients with increase in Oral Nitric Oxide levels | one year
  To determine if oral NO correlates to activity of disease in EoE

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials